CLINICAL TRIAL: NCT00905827
Title: Patient and Provider Outcomes of E-Learning Training in Collaborative Assessment and Management of Suicidality
Acronym: CAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Medical University of South Carolina (Other); Washington Psychological Center (Unknown)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EDU 08-424; 19016 (Other: MUSC IRB)
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-10

CONDITIONS: Suicide
Keywords: suicide; assessment; management; Provider Training; health services
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention 1: in person CAMS (Experimental): In person Collaborative Assessment and Management of Suicidality (CAMS) training for providers
  Interventions: Behavioral: CAMS
- Intervention 2: e-learning CAMS (Experimental): Online Collaborative Assessment and Management of Suicidality (CAMS) training for providers
  Interventions: Behavioral: CAMS
- Control: no training (No Intervention): Control Group: no training

INTERVENTIONS:
Behavioral: CAMS — Collaborative assessment management in suicidality
  Arms: Intervention 1: in person CAMS; Intervention 2: e-learning CAMS

SUMMARY:
Suicide prevention among military Veterans has become a national priority; yet, there is a gap in suicide-specific intervention training for mental health students and professionals. The need for training in this area has become even more acute with the recent hiring by the Veterans Health Affairs (VHA) of thousands of clinicians to address the mental health needs of Veterans from all war eras. Since e-learning (online) education is more effective than traditional in-person (face-to-face) education for adult learners when methods, such as blended learning, are used, this mode of delivery may more easily meet the training and continuing education needs of busy medical professionals who may find it easier to fit online education into their daily schedules.

A well developed in-person training approach known as the Collaborative Assessment and Management of Suicidality (or CAMS) has been recommended in systematic reviews as an effective tool for assessing and managing suicidality, as well as decreasing providers' fears, improving their attitudes, increasing their knowledge, confidence, and competence, and dispelling myths. The overall aims of this project were to develop an e-learning alternative for the CAMS program, determine its effectiveness relative to in-person CAMS training, and assess factors that may relate to adoption and implementation of CAMS in general and specifically through e-learning and in-person modalities.

DETAILED DESCRIPTION:
There were four specific aims:

1. Refine a Collaborative Assessment and Management of Suicidality (or CAMS) e-learning course that covers the same material and meets the same learning objectives of CAMS in-person training.
2. Test the effectiveness of the CAMS e-learning modality compared to the CAMS in-person modality and a concurrent non-intervention control in terms of provider evaluation and behavior.

   HO: Providers in each of the two CAMS arms will demonstrate higher levels of content mastery and confidence in acquired skills than providers in the no CAMS arm.

   H2: In the 12 months post-training, suicidal patients of providers in each of the two CAMS arms will receive higher rates of CAMS guideline concordant treatment, compared with providers in the no CAMS arm.
3. Test the effectiveness of the CAMS e-Learning delivery compared to the CAMS in-person delivery and a concurrent non-intervention control in terms of patient outcomes.

   H3, 4, 5: In the 12 months post-training, suicidal patients of CAMS e-learning providers and CAMS in-person providers will be similar for health services use patterns, duration of high risk episodes, and number of high risk episodes per patient.

   H6: In the 12 months post training, suicidal patients of providers in the no CAMS arm will have higher rates of emergency room use and inpatient mental health admissions, have a longer average duration of high risk episodes, and have more high risk episodes per patient.
4. Assess factors that facilitate or inhibit adoption of CAMS through e-Learning or In-person.

Of the 309 providers who met eligibility criteria, 230 consented and 212 completed the baseline assessments and were randomized. A total of 261 patients met eligibility criteria and information was abstracted on them.

We developed the CAMS-e, conducted a pilot, revised the e-CAMS, delivered the training in the first site, and again revised it. There is little difference in satisfaction ratings between the two types of training deliveries on the VA Evaluation of Training. Findings show that there were some modest immediate improvements due to the two training conditions; however, the effects were only sustainable at three months for one question related to hospitalization beliefs.

To date, the project has had the following impacts:

1. success in obtaining 6.5 continuing education units (CEUs) for the e-learning version
2. invitations to place e-CAMS on the Department of Defense learning platforms
3. VA Central Office has purchased a license to use the Suicide Status Form (SSF) as a clinical tool and template in the computerized electronic patient record system throughout the national VA. The template is in the developmental process.
4. Efforts are underway to move the CAMS e-learning on to the VA Training Management System (TMS) which will facilitate system wide dissemination and has the potential to increase adoption in VAMC's or by providers.

Additional impacts may be evident with regard to improved care once we complete analysis of the patient outcomes and provider adherence data. We have also considered a short manuscript on economic analysis

ELIGIBILITY:
Inclusion Criteria:

* Mental health providers, psychiatrist, social workers, psychologist, advanced practice nurses and case managers

Exclusion Criteria:

* Previous CAMS Training

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M. Magruder, PhD MPH BA, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (5):
- United States (5):
  - VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - VA Medical Center, Tuscaloosa, Tuscaloosa, Alabama
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Wm. Jennings Bryan Dorn VA Medical Center, Columbia SC, Columbia, South Carolina

REFERENCES:
- [Result] Pearson GS, Evans LK, Hines-Martin VP, Yearwood EL, York JA, Kane CF. Promoting the mental health of families. Nurs Outlook. 2014 May-Jun;62(3):225-7. doi: 10.1016/j.outlook.2014.04.003. No abstract available. PMID 24959633
- [Result] Puntil C, York J, Limandri B, Greene P, Arauz E, Hobbs D. Competency-based training for PMH nurse generalists: inpatient intervention and prevention of suicide. J Am Psychiatr Nurses Assoc. 2013 Jul-Aug;19(4):205-10. doi: 10.1177/1078390313496275. PMID 23950543
- [Result] Marshall E, York J, Magruder K, Yeager D, Knapp R, De Santis ML, Burriss L, Mauldin M, Sulkowski S, Pope C, Jobes DA. Implementation of online suicide-specific training for VA providers. Acad Psychiatry. 2014 Oct;38(5):566-74. doi: 10.1007/s40596-014-0039-5. Epub 2014 Feb 22. PMID 24563240
- [Result] York JA, Lamis DA, Pope CA, Egede LE. Veteran-specific suicide prevention. Psychiatr Q. 2013 Jun;84(2):219-38. doi: 10.1007/s11126-012-9241-3. PMID 23011459

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention 1: In-person CAMS: Intervention: in-person CAMS training
- Intervention 2: E-learning CAMS: Intervention: e-learning CAMS training
- Control: Control: no training
Period: Overall Study
Arm/Group | Intervention 1: In-person CAMS | Intervention 2: E-learning CAMS | Control
Started | 70 | 69 | 73
Completed | 70 | 69 | 73
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: comparison of three arms
Groups:
- Intervention 1: In-person CAMS: Intervention: in-person CAMS training for providers
- Intervention: E-training CAMS: Intervention: e-training CAMS training for providers
- Total: Total of all reporting groups
Arm/Group | Intervention 1: In-person CAMS | Intervention: E-training CAMS | Control | Total
Number analyzed (Participants) | 70 | 69 | 73 | 212
Age, Customized [Number; unit: participants]
  20-29 years | 4 | 4 | 6 | 14
  30-39 years | 22 | 22 | 23 | 67
  40-49 years | 15 | 13 | 22 | 50
  50-59 years | 19 | 22 | 18 | 59
  60-69 years | 10 | 8 | 4 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 49 | 59 | 155
  Male | 23 | 20 | 14 | 57
Race/Ethnicity, Customized [Number; unit: participants] — Not all participants reported race, hence there may be differences in overall number
  participants
    White | 45 | 45 | 46 | 136
    African American | 15 | 19 | 14 | 48
    Hispanic | 0 | 2 | 1 | 3
    Other | 6 | 1 | 4 | 11
Profession [Number; unit: participants]
  Psychiatrist | 12 | 12 | 12 | 36
  Psychologist | 16 | 13 | 18 | 47
  Midlevel Provider | 42 | 44 | 43 | 129

OUTCOME MEASURES:

1. Primary Outcome: Provider Self-efficacy and Beliefs About Suicidality
Description: Assessed beliefs and confidence in managing suicidal individuals. Using a 5-point Likert scale, there were 11 items that addressed the following: competence, reactions, beliefs, motivations, and CAMS as it relates to their practice. Scores ranged from 11-55 with questions were phrased so higher scores indicated more positive views.
Time Frame: post-training
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention 1: In-person CAMS | Intervention 2: E-learning CAMS | Control
Number analyzed (Participants) | 70 | 69 | 73
units on a scale | 45.6 (0.5) | 44.9 (0.5) | 43.0 (0.6)
Statistical Analysis 1: Comparison: Intervention 1: In-person CAMS vs Control; Pairwise comparisons (ANOVA simple effect comparisons) adjusted for baseline scores; Test type: Superiority or Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Intervention 2: E-learning CAMS vs Control; Pairwise comparisons (ANOVA simple effect comparisons) adjusted for baseline scores; Test type: Superiority or Other; p = 0.01, ANOVA

2. Secondary Outcome: Satisfaction With Training
Description: Evaluation included 20 standard items assessing providers satisfaction with training, including items similar to other published satisfaction surveys. Survey items were rated using a five-point Likert scale indicating the degree to which respondents agreed or disagreed. Questions were always phrased positively so that agree or strongly agree is equivalent to a positive response.
Time Frame: post-training
Measure: Number; unit: participants
Arm/Group | Intervention 1: In-person CAMS | Intervention 2: E-learning CAMS
Number analyzed (Participants) | 70 | 69
participants
  Agree | 66 | 62
  Neutral | 3 | 2
  Disagree | 1 | 5

ADVERSE EVENTS:
Time Frame: 1 year
Description: DSMB assembled annually
Groups:
- Arm 1: Intervention: in person CAMS training for providers
  CAMS: Collaborative assessment management in suicidality
- Arm 2: Intervention: e-learning CAMS training for providers
  CAMS: Collaborative assessment management in suicidality
- Arm 3: Control Group: no training
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/69 | 0/73
Other Adverse Events (participants affected / at risk) | 0/70 | 0/69 | 0/73

LIMITATIONS AND CAVEATS:
Providers in this VISN may not be representative of providers in other VAMCs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes